CLINICAL TRIAL: NCT00028795
Title: A Phase II Study of Temozolomide in the Treatment of Children With High Grade Glioma
Brief Title: Chemotherapy and Radiation Therapy After Surgery in Treating Children With Newly Diagnosed Astrocytoma, Glioblastoma Multiforme, Gliosarcoma, or Diffuse Intrinsic Pontine Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACNS0126; COG-ACNS0126 (Other: Children's Oncology Group); CDR0000069135 (Other: Clinical Trials.gov)
Record Dates: First submitted 2002-01-04; First posted 2003-01-27 (Estimated); Last update posted 2014-02-21 (Estimated); Status verified 2014-02

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: childhood brain stem glioma; childhood high-grade cerebral astrocytoma; childhood spinal cord neoplasm; untreated childhood brain stem glioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Astrocytoma; Spinal Cord Neoplasms | interventions — Temozolomide; Chemotherapy, Adjuvant; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemoradiotherapy (Experimental)
  Interventions: Drug: temozolomide; Procedure: adjuvant therapy; Radiation: radiation therapy

INTERVENTIONS:
Drug: temozolomide
Procedure: adjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Giving chemotherapy together with radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving chemotherapy together with radiation therapy after surgery followed by chemotherapy alone works in children with newly diagnosed astrocytoma, glioblastoma multiforme, gliosarcoma, or diffuse intrinsic pontine glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the event-free survival of patients with newly diagnosed anaplastic astrocytoma, glioblastoma multiforme, gliosarcoma, or diffuse intrinsic pontine glioma (DIPG) treated with adjuvant temozolomide administered concurrently with postoperative radiotherapy and then alone as maintenance therapy vs historical control cohorts treated in prior Pediatric Oncology Group and Children's Cancer Group studies.
* Determine the toxicity of this regimen in these patients.
* Determine the efficacy of this regimen in patients with DIPG.
* Determine the toxicity of this regimen in patients with DIPG.

OUTLINE: This is a multicenter study.

* Adjuvant chemoradiotherapy: Beginning within 6 weeks after surgical resection or diagnosis*, patients without gross residual disease undergo cranial irradiation 5 days a week for 6 weeks. Beginning within 6 weeks after surgical resection, patients with gross residual disease undergo radiotherapy as above followed by boost radiotherapy for 1 week. All patients receive oral temozolomide once daily beginning within 5 days after initiation of radiotherapy and continuing for a total of 6 weeks in the absence of disease progression or unacceptable toxicity.
* Adjuvant maintenance therapy: Beginning 4 weeks after completion of adjuvant chemoradiotherapy, patients receive oral temozolomide on days 1-5. Treatment repeats every 28 days for a total of 10 courses in the absence of disease progression or unacceptable toxicity.

NOTE: *For patients with diffuse intrinsic pontine glioma only

Patients are followed every 3-6 months for 4 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 50-60 patients will be accrued for this study within 12-14 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed newly diagnosed CNS tumor of the following types:

  * High grade glioma (HGG) of one of the following histologies:

    * Anaplastic astrocytoma (grade III)
    * Glioblastoma multiforme (grade IV)
    * Gliosarcoma
    * Primary spinal cord malignant glioma
  * Diffuse intrinsic pontine glioma (DIPG)

    * Diagnosed by gadolinium-enhanced MRI
    * At least 2/3 of tumor situated in the pons AND tumor clearly originated in the pons
    * No diffuse leptomeningeal disease
    * No tumors with features not typical of diffuse intrinsic brainstem glioma, including any of the following:

      * Dorsally exophytic brainstem glioma
      * Cervico-medullary junction tumor
      * Focal low-grade glioma of the midbrain or brainstem
    * No diffuse brainstem enlargement due to neurofibromatosis
* No primary brain stem malignant glioma
* No M+ disease (CSF positive for tumor or metastatic disease)
* Must begin study radiotherapy within 6 weeks after surgical resection (for HGG patients) or diagnosis (for DIPG patients)

PATIENT CHARACTERISTICS:

Age:

* 3 to 21

Performance status:

* Karnofsky 50-100% OR
* Lansky 50-100%

Life expectancy:

* At least 2 months

Hematopoietic:

* Absolute neutrophil count at least 1,000/mm^3
* Platelet count at least 100,000/mm^3*
* Hemoglobin at least 10.0 g/dL* NOTE: *Transfusion independent

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT or SGPT less than 2.5 times ULN

Renal:

* Creatinine no greater than 1.5 times ULN

Other:

* No other concurrent malignancy
* Concurrent seizure disorder allowed if well controlled on anticonvulsants
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 2 months after completion of study treatment

PRIOR CONCURRENT THERAPY:

Biologic:

* No concurrent routine cytokine support

Chemotherapy:

* Not specified

Endocrine therapy:

* No concurrent corticosteroids except for increased intracranial pressure in patients with CNS tumors

Radiotherapy:

* See Disease Characteristics

Surgery:

* See Disease Characteristics

Other:

* No prior therapy for HGG or DIPG

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 170 (Actual)
Dates: Start 2002-12; Primary Completion 2007-09 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Improved outcome
Toxicity as assessed by NCI CTCAE v. 2.0

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth J. Cohen, MD, MBA, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (230):
- United States (202):
  - Comprehensive Cancer Center at University of Alabama at Birmingham, Birmingham, Alabama
  - University of South Alabama Cancer Research Institute, Mobile, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Jonathan Jaques Children's Cancer Center at Miller Children's Hospital, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Samuel Oschin Comprehensive Cancer Institute at Cedars-Sinai Medical Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Medical Center, Orange, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital at Stanford University Medical Center, Palo Alto, California
  - Sutter Cancer Center, Sacramento, California
  - University of California Davis Cancer Center, Sacramento, California
  - Kaiser Permanente Medical Center - Sacramento, Sacramento, California
  - Kaiser Permanente Medical Center/Kaiser Foundation Hospital - San Diego, San Diego, California
  - Children's Hospital and Health Center - San Diego, San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Kaiser Permanente Medical Center - Santa Clara Kiely Campus, Santa Clara, California
  - General Robert Huyser Cancer Center at David Grant Medical Center, Travis Air Force Base, California
  - Children's Hospital Cancer Center, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - Carole and Ray Neag Comprehensive Cancer Center at the University of Connecticut Health Center, Farmington, Connecticut
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Lombardi Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Children's Hospital of Southwest Florida, Fort Myers, Florida
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Joe DiMaggio Children's Hospital at Memorial, Hollywood, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - Jackson Memorial Hospital, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - Baptist-South Miami Regional Cancer Program, Miami, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Nemours Children's Clinic-Orlando, Orlando, Florida
  - Sacred Heart Children's Hospital, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - St. Joseph's Children's Hospital of Tampa, Tampa, Florida
  - Kaplan Cancer Center at St. Mary's Medical Center, West Palm Beach, Florida
  - AFLAC Cancer Center and Blood Disorders Service of Children's Healthcare of Atlanta - Scottish Rite Campus, Atlanta, Georgia
  - MBCCOP-Medical College of Georgia Cancer Center, Augusta, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Curtis & Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - St. Luke's Mountain States Tumor Institute - Boise, Boise, Idaho
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois Medical Center, Chicago, Illinois
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Advocate Hope Children's Hospital, Oak Lawn, Illinois
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Children Cancer Center at Riley Hospital for Children, Indianapolis, Indiana
  - St. Vincent Hospitals and Health Care Centers, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Wesley Medical Center, Wichita, Kansas
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane Cancer Center at Tulane University Hospital and Clinic, New Orleans, Louisiana
  - Children's Hospital of New Orleans, New Orleans, Louisiana
  - Ochsner Cancer Institute at Ochsner Clinic Foundation, New Orleans, Louisiana
  - Pediatric Specialty Clinic at Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Alvin and Lois Lapidus Cancer Institute at Sinai Hospital, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Walter Reed Army Medical Center, Silver Spring, Maryland
  - Floating Hospital for Children, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Baystate Regional Cancer Program at D'Amour Center for Cancer Care, Springfield, Massachusetts
  - UMASS Memorial Cancer Center - University Campus, Worcester, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, Lansing, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - St. Mary's - Duluth Clinic Cancer Center, Duluth, Minnesota
  - Children's Hospitals and Clinics - Minneapolis/St. Paul, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri - Columbia, Columbia, Missouri
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - St. Louis Children's Hospital, St Louis, Missouri
  - Children's Hospital of Omaha, Omaha, Nebraska
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - Valerie Fund Children's Center at Atlantic Health, Summit, New Jersey
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - Children's Hospital at Albany Medical Center, Albany, New York
  - Brooklyn Hospital Center, Brooklyn, New York
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Brookdale University Hospital and Medical Center, Brooklyn, New York
  - Comprehensive Cancer Center at Maimonides Medical Center, Brooklyn, New York
  - Schneider Children's Hospital, New Hyde Park, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Long Island Cancer Center at Stony Brook University Hospital, Stony Brook, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Leo W. Jenkins Cancer Center at Pitt County Memorial Hospital, Greenville, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Dakota Cancer Institute at Innovis Health - Dakota Clinic, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Ireland Cancer Center at University Hospitals of Cleveland and Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Columbus Children's Hospital, Columbus, Ohio
  - Children's Medical Center - Dayton, Dayton, Ohio
  - Toledo Children's Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Tod Children's Hospital - Forum Health, Youngstown, Ohio
  - Children's Hospital at Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center & Children's Hospital, Portland, Oregon
  - Doernbecher Children's Hospital at Oregon Health & Science University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Palmetto Health South Carolina Cancer Center, Columbia, South Carolina
  - Children's Hospital of Greenville Hospital System, Greenville, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota
  - East Tennessee State University Cancer Center at Johnson City Medical Center, Johnson City, Tennessee
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - Texas Tech University Health Sciences Center School of Medicine, Amarillo, Texas
  - Children's Hospital of Austin, Austin, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Simmons Cancer Center at University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - M.D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - San Antonio Military Pediatric Cancer and Blood Disorders Center, Lackland Air Force Base, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - MBCCOP - South Texas Pediatrics, San Antonio, Texas
  - Methodist Cancer Center at Methodist Specialty and Transplant Hospital, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Center for Cancer Prevention and Care at Scott and White Clinic, Temple, Texas
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - Vermont Cancer Center at University of Vermont, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - INOVA Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Massey Cancer Center at Virginia Commonwealth University, Richmond, Virginia
  - Carilion Medical Center for Children at Roanoke Community Hospital, Roanoke, Virginia
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Deaconess Medical Center, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center - Tacoma, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University - Robert C. Byrd Health Sciences Center - Charleston Division, Charleston, West Virginia
  - Cabell Huntington Hospital, Huntington, West Virginia
  - Mary Babb Randolph Cancer Center at West Virginia University Hospitals, Morgantown, West Virginia
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (6):
  - Sydney Children's Hospital, Randwick, New South Wales
  - Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Children's Hospital, Brisbane, Queensland
  - Women's and Children's Hospital, North Adelaide, South Australia
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (15):
  - Alberta Children's Hospital, Calgary, Alberta
  - Cross Cancer Institute at University of Alberta, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Children's Health and Rehabilitation Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Children's Hospital of Western Ontario, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Montreal Children's Hospital at McGill University Health Center, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
  - Centre de Recherche du Centre Hospitalier de l'Universite Laval, Sainte-Foy, Quebec
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- University Medical Center Groningen, Groningen, Netherlands
- Starship Children's Health, Auckland, New Zealand
- Puerto Rico (2):
  - Puerto Rico Cancer Center at University of Puerto Rico - Medical Sciences Campus, San Juan
  - San Jorge Children's Hospital, Santurce
- Switzerland (3):
  - Swiss Pediatric Oncology Group Bern, Bern
  - Swiss Pediatric Oncology Group Geneva, Geneva
  - Swiss Pediatric Oncology Group Lausanne, Lausanne

REFERENCES:
- [Background] Pollack IF, Hamilton RL, Burger PC, Brat DJ, Rosenblum MK, Murdoch GH, Nikiforova MN, Holmes EJ, Zhou T, Cohen KJ, Jakacki RI; Children's Oncology Group. Akt activation is a common event in pediatric malignant gliomas and a potential adverse prognostic marker: a report from the Children's Oncology Group. J Neurooncol. 2010 Sep;99(2):155-63. doi: 10.1007/s11060-010-0297-3. Epub 2010 Jul 4. PMID 20607350
- [Background] Pollack IF, Hamilton RL, Sobol RW, Nikiforova MN, Nikiforov YE, Lyons-Weiler MA, LaFramboise WA, Burger PC, Brat DJ, Rosenblum MK, Gilles FH, Yates AJ, Zhou T, Cohen KJ, Finlay JL, Jakacki RI; Children's Oncology Group. Mismatch repair deficiency is an uncommon mechanism of alkylator resistance in pediatric malignant gliomas: a report from the Children's Oncology Group. Pediatr Blood Cancer. 2010 Dec 1;55(6):1066-71. doi: 10.1002/pbc.22634. PMID 20589656
- [Result] Cohen KJ, Heideman RL, Zhou T, Holmes EJ, Lavey RS, Bouffet E, Pollack IF. Temozolomide in the treatment of children with newly diagnosed diffuse intrinsic pontine gliomas: a report from the Children's Oncology Group. Neuro Oncol. 2011 Apr;13(4):410-6. doi: 10.1093/neuonc/noq205. Epub 2011 Feb 22. PMID 21345842
- [Result] Cohen KJ, Pollack IF, Zhou T, Buxton A, Holmes EJ, Burger PC, Brat DJ, Rosenblum MK, Hamilton RL, Lavey RS, Heideman RL. Temozolomide in the treatment of high-grade gliomas in children: a report from the Children's Oncology Group. Neuro Oncol. 2011 Mar;13(3):317-23. doi: 10.1093/neuonc/noq191. PMID 21339192
- [Result] Nicholson HS, Kretschmar CS, Krailo M, Bernstein M, Kadota R, Fort D, Friedman H, Harris MB, Tedeschi-Blok N, Mazewski C, Sato J, Reaman GH. Phase 2 study of temozolomide in children and adolescents with recurrent central nervous system tumors: a report from the Children's Oncology Group. Cancer. 2007 Oct 1;110(7):1542-50. doi: 10.1002/cncr.22961. PMID 17705175